CLINICAL TRIAL: NCT03344887
Title: An Innovative Trial Assessing Donor Sex on Recipient Mortality (iTADS)
Brief Title: An Innovative Trial Assessing Donor Sex on Recipient Mortality
Acronym: iTADS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Blood Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20170477-01H
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Red Blood Cell Transfusion
Keywords: anemia; donor sex; prospective blinded pragmatic randomized
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RBC Transfusion from male donor (Active Comparator): For the treatment of anemia
  Interventions: Other: RBC Transfusion from male donor
- RBC Transfusion from female donor (Active Comparator): For the treatment of anemia
  Interventions: Other: RBC Transfusion from female donor

INTERVENTIONS:
Other: RBC Transfusion from male donor — Patients requiring an RBC transfusion for the treatment of anemia will receive products from a male donor at initial and any subsequent hospitalizations during the trial period.
  Arms: RBC Transfusion from male donor
Other: RBC Transfusion from female donor — Patients requiring an RBC transfusion for the treatment of anemia will receive products from a female donor at initial and any subsequent hospitalizations during the trial period.
  Arms: RBC Transfusion from female donor

SUMMARY:
The iTADS trial will test an important blood donor characteristic - donor sex - to see whether male donor blood leads to a greater benefit for transfusion recipients compared to female donor blood.

The trial will help determine how the investigators can tailor the selection of blood donors based on donor characteristics (e.g. sex) to further improve the safety and optimize the clinical benefit of blood products in Canada.

DETAILED DESCRIPTION:
The investigators have designed an innovative pragmatic randomized trial that will allocate transfusion recipients to receive either only male or only female donor transfusions.

Primary objective:

To confirm that a transfusion strategy of receiving male donor RBC (Red Blood Cell) units only will improve survival compared to a transfusion strategy of female donor RBC units in all hospital patients requiring a transfusion.

Secondary objectives:

1. To assess effects of male RBC units on major morbidities (cancer, infection, end-organ damage)
2. To assess effects across major patient subgroups (major surgery, intensive care, oncology)
3. To assess the effect of female donor pregnancy history on recipient transfusion outcome
4. To build capacity to conduct large innovative prospective pragmatic clinical trials in transfusion medicine using routinely collected clinical and administrative information.

ELIGIBILITY:
Inclusion Criteria:

* All patients (excluding neonates) requiring one or more allogeneic RBC transfusions for the treatment of anemia will be included.

Exclusion Criteria:

* Patients that do not have a valid Ontario Health Insurance Plan (OHIP) number at time of first transfusion
* Patients that require emergent release of a RBC transfusion and in whom emergency randomization could not be completed
* Patients with complex antibody profile in which it is impossible to match RBC units

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8850 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2021-01-23 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 2 years
  Measured from date of first randomization to date of death or end of study 2 years from first patient enrollment.

SECONDARY OUTCOMES:
Survival | 30 days, 3 months, 6 months and 1 year
  Measured from date of first randomization to date of death or end of study 2 years from the first patient enrollment.
Length of hospital stay | 2 years
  Number of days admitted to hospital for the treatment of anemia.
New ICU admission | 2 years
  Occurrence of ICU admission(s) once discharged for the treatment of anemia.
Re-hospitalization | 2 years
  Occurrence of additional hospital admission(s) once discharged for the treatment of anemia.
Health system costs | 2 years
  The cost of the treatment of anemia and any related downstream health care resources.
Occurrence of new cancer | 2 years
  The number of new cancer diagnoses, not present during the initial treatment of anemia.
Recurrence of cancer | 2 years
  The number of repeat cancer diagnoses, diagnosed previous to the initial treatment of anemia.
Infection rates | 2 years
  Methicillin-resistant Staphylococcus aureus and Clostridium difficile for hospital-acquired infections.
New occurrence of hemodialysis | 2 years
  For severe chronic renal failure.
Myocardial infarctions | 2 years
  For cardiac events.

CONTACTS AND LOCATIONS:
Overall Officials: Michaël Chassé, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Dean Fergusson, Principal Investigator — Ottawa Hospital Research Institute; Alan Tinmouth, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital - General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chasse M, Fergusson DA, Tinmouth A, Acker JP, Perelman I, Tuttle A, English SW, Hawken S, Forster AJ, Shehata N, Thavorn K, Wilson K, Cober N, Maddison H, Tokessy M. Effect of Donor Sex on Recipient Mortality in Transfusion. N Engl J Med. 2023 Apr 13;388(15):1386-1395. doi: 10.1056/NEJMoa2211523. PMID 37043654
- [Derived] Fergusson DA, Chasse M, Tinmouth A, Acker JP, English S, Forster AJ, Hawken S, Shehata N, Thavorn K, Wilson K, Tuttle A, Perelman I, Cober N, Maddison H, Tokessy M. Pragmatic, double-blind, randomised trial evaluating the impact of red blood cell donor sex on recipient mortality in an academic hospital population: the innovative Trial Assessing Donor Sex (iTADS) protocol. BMJ Open. 2021 Feb 23;11(2):e049598. doi: 10.1136/bmjopen-2021-049598. PMID 33622960